CLINICAL TRIAL: NCT06734273
Title: Randomized Control Trial of Sleeve Gastrectomy with Tirzepatide in Maximizing Weight Loss
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nicholas Skertich (Other)
Responsible Party: Sponsor-Investigator, Nicholas Skertich, Assistant Professor, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24101008
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SG-T: sleeve gastrectomy with tirzepatide (Experimental): In this study, the intervention group (n=21) are patients who will undergo sleeve gastrectomy and receive tirzepatide. Patients who were selected in this arm will undergo a 4-week dose escalation period. Starting at 6 months after surgery they will receive weekly 2.5mg doses (for 4 weeks). Afterwards, they will receive weekly 5mg doses. They will maintain this dose until 12 months after surgery.
  Interventions: Drug: Mounjaro; Procedure: Sleeve Gastrectomy
- SG-A: sleeve gastrectomy alone (Active Comparator): In this study the control group (n=21) are patients who will undergo sleeve gastrectomy alone.
  Interventions: Procedure: Sleeve Gastrectomy

INTERVENTIONS:
Drug: Mounjaro — In this study, the intervention group (n=21) are patients who will undergo sleeve gastrectomy and receive tirzepatide after surgery. Patients who were selected in this arm will undergo a 4-week dose escalation period. Starting at 6 months they will receive weekly 2.5mg doses (for 4 weeks). Afterwards, they will receive weekly 5mg doses. They will maintain this dose until 12 months after surgery.
  Arms: SG-T: sleeve gastrectomy with tirzepatide
Procedure: Sleeve Gastrectomy — Subjects in both the interventional group (n=21) and the control group (n=21) will undergo sleeve gastrectomy.

SUMMARY:
This study examines whether adding tirzepatide-a medication that helps with weight loss-after sleeve gastrectomy surgery can help people lose more weight after the surgery; better improve conditions like Type 2 diabetes, high blood pressure, high cholesterol, and sleep apnea after surgery and; whether this causes more complications or side effects compared to surgery alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 to 65 years of age
* Body Mass Index >35 with comorbidity of Type 2 Diabetes and/or Hypertension and/or Hyperlipidemia and/or Obstructive Sleep Apnea OR Body Mass Index >40 with or without comorbidity
* Undergoing primary sleeve gastrectomy

Exclusion Criteria:

* Prior metabolic and bariatric surgery
* Prior use of GLP-1 agonist
* Prior history of pancreatitis
* Personal/family history of medullary thyroid cancer or MEN type 2
* Secondary cause of obesity
* Any eating disorder
* Pregnancy/lactation
* History of acute coronary syndrome or myocardial infarction
* History of stroke
* Hepatic dysfunction: AST/ALT >3 ULN
* Renal dysfunction eGFR<45ml/min/1.73m2
* Active malignancy
* History of diabetic retinopathy
* History of gastroparesis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 12 months after surgery

SECONDARY OUTCOMES:
Weight Loss | 18 months after surgery
Type 2 Diabetes | 12 months after surgery
  Researchers will use Hemoglobin A1c (%) to measure Type 2 Diabetes. A lower value indicates improvement.
Type 2 Diabetes | 18 months after surgery
  Researchers will use Hemoglobin A1c (%) to measure Type 2 Diabetes. A lower value indicates improvement.
High Blood Pressure | 12 months after surgery
High Blood Pressure | 18 months after surgery
High Cholesterol | 12 months after surgery
  Researchers will measure Cholesterol by the number of cholesterol-lowering medications needed by the subject (#). A lower value indicates improvement.
High Cholesterol | 18 months after surgery
  Researchers will measure Cholesterol by the number of cholesterol-lowering medications needed by the subject (#). A lower value indicates improvement.
Sleep Apnea | 12 months after surgery
  Researchers will measure Sleep Apnea by subject's need for a CPAP (continuous positive airway pressure) machine (Y/N).
Sleep Apnea | 18 months after surgery
  Researchers will measure Sleep Apnea by subject's need for a CPAP (continuous positive airway pressure) machine (Y/N)
Complications/Side Effects | 12 months after surgery
Complications/Side Effects | 18 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Skertich, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results will be made available following publication for a period of 3 years, dependent on IRB approval to share the data and execution of a data use agreement. Access will be granted to researchers who submit a methodologically sound proposal approved by their IRB. Requests for data access can be made to the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start: after publication. End: 3 years after publication.
Access Criteria: De-identified individual participant data (IPD) that underlie the results will be made available following publication for a period of 3 years, dependent on IRB approval to share the data and execution of a data use agreement. Access will be granted to researchers who submit a methodologically sound proposal approved by their IRB. Requests for data access can be made to the Principal Investigator.